CLINICAL TRIAL: NCT00811577
Title: A Phase 2a Double Blind, Placebo Within-Patient Controlled, Multi-Center Dose Ranging Study to Evaluate the Safety and Preliminary Efficacy of AZX100 Drug Product in Trocar Sites of Arthroscopic Shoulder Surgery Patients
Brief Title: A Phase 2a Study to Evaluate the Safety and Efficacy of AZX100 in Trocar Sites of Arthroscopic Shoulder Surgery Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capstone Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OL-ASCAR-03
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2012-10-11 (Estimated); Status verified 2012-09

CONDITIONS: Scar Prevention; Scar Reduction
Keywords: AZX100; Patient and Observer Scar Assessment Scale; POSAS; Visual Analog Scale; VAS; Trocar; Scarring; Scar reduction; Scar prevention
MeSH Terms: conditions — Cicatrix | interventions — AZX 100

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZX100-placebo (Experimental): Three trocar sites designated as anterior, lateral and posterior were randomized on each patient to receive one low dose of AZX100 3 mg/linear cm, one high dose of AZX100 10 mg/linear cm, or placebo (saline).
  Interventions: Drug: Placebo; Drug: AZX100
- Placebo-only (Placebo Comparator): Three trocar sites on each patient received one dose of placebo (saline).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Patients in the Placebo-only arm were dosed intradermally with placebo (saline) in three trocar sites on Day 9 (plus/minus 2 days) and Day 21 (plus/minus 2 days) after arthroscopic shoulder surgery. In the AZX100-placebo arm, 3 or 10 mg or placebo (saline) was administered intradermally at each of three trocar sites on each patient 9 ± 2 days and 21 ± 2 days after arthroscopic surgery. The three trocar sites (anterior, lateral, and posterior sides of the shoulder) were randomized to receive the same dose of study agent for both dose administrations.
Drug: AZX100 — AZX100 Drug Product 3 or 10 mg or placebo (saline) was administered intradermally at each of three trocar sites on each patient 9 ± 2 days and 21 ± 2 days after arthroscopic surgery. The three trocar sites (anterior, lateral, and posterior sides of the shoulder) were randomized to receive the same dose of study agent for both dose administrations.
  Arms: AZX100-placebo

SUMMARY:
The purpose of this study was to determine the safety of AZX100 Drug Product and to determine whether it was effective in preventing or reducing scars that were made from trocars following arthroscopic shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for an arthroscopic shoulder surgery that will result in at least 3 trocar sites
* Healthy male or non-pregnant female 18-75 years old
* Non-diabetic
* Body Mass Index 18-35
* No clinically significant abnormal values on blood test
* Non-smoker for previous 6 months

Exclusion Criteria:

* History of acute or chronic disease
* Cancer within previous 5 years, except for removed skin cancer
* Hypersensitivity reaction
* Allergy to general anesthesia, lidocaine, or epinephrine
* Current skin disorder other than folliculitis or acne
* On therapy with steroids
* On therapy with a drug that affects collagen synthesis
* Positive for HIV or hepatitis
* Positive urine test for nicotine
* Positive blood test for anti-AZX100 antibodies
* Participated in another clinical study within 60 days before enrollment
* Gave blood within 7 days before dosing
* Gave plasma within 3 days before dosing
* Tattoo on the shoulder area
* Applied any prescribed or over the counter agents to the shoulder within 14 days before dosing, or intend to use any scar improving product
* Visited a tanning salon within 14 days before dosing
* History of drug addiction or excessive use of alcohol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Lotus Clinical Research, Inc., Pasadena, California
  - Florida Research Associates, DeLand, Florida
  - Atlas Orthopedics & Sports Medicine, Orlando, Florida
  - Orthopaedics East, PA, Greenville, North Carolina
  - Texas Orthopedics, Sports & Rehab Assoc., Austin, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment in the study began in January 2009 and was completed in December 2009. All patients were enrolled in dermatological medical clinics.
Groups:
- AZX100-Placebo Arm: Three trocar sites designated as anterior, lateral and posterior will be randomized on each patient to receive one low dose of AZX100, one high dose of AZX100, or placebo.
- Placebo-only Arm: Three trocar sites on each patient will receive one dose of placebo.
Period: Overall Study
Arm/Group | AZX100-Placebo Arm | Placebo-only Arm
Started | 126 | 24
Completed | 116 | 23
Not Completed | 10 | 1
Not completed — Lost to Follow-up | 7 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZX100-Placebo Arm | Placebo-only Arm | Total
Number analyzed (Participants) | 126 | 24 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 112 | 19 | 131
  >=65 years | 14 | 5 | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 51.3 (11.8) | 51.8 (13.2) | 51.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 7 | 43
  Male | 90 | 17 | 107
Region of Enrollment [Number; unit: participants]
  United States | 126 | 24 | 150

OUTCOME MEASURES:

1. Primary Outcome: Differences Among the 3 Dosage Groups in the Patient (PSAS) and Observer (OSAS) Scar Assessment Scale (POSAS) Scores
Description: Efficacy was based on the difference between mean POSAS scores of placebo and 3 mg AZX100, and placebo and 10 mg AZX100 12 months after shoulder surgery. Three trocar sites were randomized on each patient to receive AZX100 3 mg or AZX100 10 mg or placebo at 9 days and 21 days after shoulder surgery. PSAS results included patients' ratings on a scale of 1-10 (1 was normal skin or no complaints and 10 was the worst imaginable scar or the worst difference) for the following: Is the scar painful? Is the scar itching? Is the color of the scar different? Is the scar more stiff? Is the thickness of the scar different? Is the scar irregular? The possible minimum score was 6 and the maximum (worst) score was 60. OSAS results included observers' ratings on a scale of 1-10 (1 was normal skin and 10 was the worst scar imaginable) for vascularization, pigmentation, thickness, relief, and pliability. The possible minimum score was 5 and the possible maximum (worst) score was 50.
Time Frame: 12 months
Population: The efficacy analysis was based on patient data from the AZX100/Placebo cohort (i.e., not including the patients receiving placebo-only). In the ITT sample for the POSAS outcomes, available sample sizes were 122 at Day 42 and 113 at Month 12 (including 4 subjects who withdrew from the study but were still followed for safety until Month 12).
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- PSAS Results for Placebo Trocar Scars: This group included PSAS results at 12 months for trocar scars that were randomized to receive saline placebo/cm at 9 days and 21 days following shoulder surgery.
- PSAS Results for 3 mg AZX100 Trocar Scars: This group included PSAS results at 12 months for trocar scars that were randomized to receive AZX100 3 mg/cm at 9 days and 21 days following shoulder surgery.
- PSAS Results for 10 mg AZX100 Trocar Scars: This group included PSAS results at 12 months for trocar scars that were randomized to receive AZX100 10 mg/cm at 9 days and 21 days following shoulder surgery.
- OSAS Results for Placebo Trocar Scars: This group included OSAS results at 12 months for trocar scars that were randomized to receive saline placebo/cm at 9 days and 21 days following shoulder surgery.
- OSAS Results for 3 mg AZX100 Trocar Scars: This group included OSAS results at 12 months for trocar scars that were randomized to receive AZX100 3 mg/cm at 9 days and 21 days following shoulder surgery.
- OSAS Results for 10 mg AZX100 Trocar Scars: This group included OSAS results at 12 months for trocar scars that were randomized to receive AZX100 10 mg/cm at 9 days and 21 days following shoulder surgery.
Arm/Group | PSAS Results for Placebo Trocar Scars | PSAS Results for 3 mg AZX100 Trocar Scars | PSAS Results for 10 mg AZX100 Trocar Scars | OSAS Results for Placebo Trocar Scars | OSAS Results for 3 mg AZX100 Trocar Scars | OSAS Results for 10 mg AZX100 Trocar Scars
Number analyzed (Participants) | 113 | 113 | 113 | 113 | 113 | 113
Units on a scale | 8.0 (4.1) | 8.0 (4.7) | 8.3 (5.0) | 6.8 (2.7) | 6.8 (2.5) | 6.9 (2.5)
Statistical Analysis 1: Comparison: PSAS Results for Placebo Trocar Scars vs PSAS Results for 3 mg AZX100 Trocar Scars; Using serial gate-keeping to preserve the 5% overall type I error of 1-4 two-sided tests, 2-sided Wilcoxon Signed Rank tests were used. Computer graphics were used to display outcomes at Month 12, compare paired differences of outcomes between the 2 dosages and placebo, and show time trends in mean outcomes. Repeated measures regression models (GEE models in SAS/STAT PROC GENMOD) were used to examine longitudinal outcomes with terms for treatment and trocar location adjusted for key covariates; Test type: Superiority or Other; p = 0.57, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 2: Comparison: PSAS Results for Placebo Trocar Scars vs PSAS Results for 10 mg AZX100 Trocar Scars; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.56, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 3: Comparison: OSAS Results for Placebo Trocar Scars vs OSAS Results for 3 mg AZX100 Trocar Scars; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.61, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 4: Comparison: OSAS Results for Placebo Trocar Scars vs OSAS Results for 10 mg AZX100 Trocar Scars; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.80, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used

2. Secondary Outcome: Between-group Mean Differences in Visual Analog Scale Scores Rated by Independent Blinded Raters Using 3D Photography
Description: Three trocar sites were randomized on each patient to receive AZX100 3 mg/cm or AZX100 10 mg/cm or saline placebo/cm at 9 days and 21 days after surgery. Twelve months after surgery, images of the trocar sites were longitudinally evaluated and rated using a standard 100 mm Visual Analog Scale (VAS) by two blinded independent dermatologists, with 0 being normal skin and 100 being the worst scar imaginable. Efficacy was based on the difference between VAS scores of placebo and 3 mg AZX100 and placebo and 10 mg AZX100 for each of the two raters separately. Data from both raters was not combined.
Time Frame: 12 months
Population: Efficacy analysis was based on patient data from the AZX100/Placebo cohort (i.e., not including patients receiving placebo-only). In the ITT sample for the VAS outcome, available sample sizes were 122 at Day 42 and 113 at Month 12 (including four subjects who withdrew from the study but were still followed for safety until Month 12).
Measure: Mean (Standard Deviation); unit: Millimeters
Groups:
- Rater 1 VAS Scores for Placebo Trocar Scars; Rater 2 VAS Scores for Placebo Trocar Scars: This group included VAS scores at the 12 month time point for trocar scars that were randomized to receive saline placebo/cm at 9 days and 21 days following shoulder surgery.
- Rater 1 VAS Scores for 3 mg AZX100 Trocar Scars; Rater 2 VAS Scores for 3 mg AZX100 Trocar Scars: This group included VAS scores at the 12 month time point for trocar scars that were randomized to receive AZX100 3 mg/cm at 9 days and 21 days following shoulder surgery.
- Rater 1 VAS Scores for 10 mg AZX100 Trocar Scars; Rater 2 VAS Scores for 10 mg AZX100 Trocar Scars: This group included VAS scores at the 12 month time point for trocar scars that were randomized to receive AZX100 10 mg/cm at 9 days and 21 days following shoulder surgery.
Arm/Group | Rater 1 VAS Scores for Placebo Trocar Scars | Rater 1 VAS Scores for 3 mg AZX100 Trocar Scars | Rater 1 VAS Scores for 10 mg AZX100 Trocar Scars | Rater 2 VAS Scores for Placebo Trocar Scars | Rater 2 VAS Scores for 3 mg AZX100 Trocar Scars | Rater 2 VAS Scores for 10 mg AZX100 Trocar Scars
Number analyzed (Participants) | 113 | 113 | 113 | 113 | 113 | 113
Millimeters | 10.96 (8.58) | 11.78 (9.91) | 11.86 (7.21) | 17.23 (12.25) | 17.49 (11.66) | 18.49 (11.20)
Statistical Analysis 1: Comparison: Rater 1 VAS Scores for Placebo Trocar Scars vs Rater 1 VAS Scores for 3 mg AZX100 Trocar Scars; Using a 100 mm VAS scale, each photograph was assessed by two raters, who, in an end-of-study session, were presented with photographs in their longitudinal sequence, but blinded as to dosage group. These data were used for an inter-rater concordance analysis and also to compare the placebo, 3 and 10 mg dosages; Test type: Superiority or Other; p = 0.47, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 2: Comparison: Rater 1 VAS Scores for Placebo Trocar Scars vs Rater 1 VAS Scores for 10 mg AZX100 Trocar Scars; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.080, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 3: Comparison: Rater 2 VAS Scores for Placebo Trocar Scars vs Rater 2 VAS Scores for 3 mg AZX100 Trocar Scars; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.96, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 4: Comparison: Rater 2 VAS Scores for Placebo Trocar Scars vs Rater 2 VAS Scores for 10 mg AZX100 Trocar Scars; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.22, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used

3. Secondary Outcome: Between-group Mean Differences in Objective Measures Via 3D Photography (Elevation, Length, Width)
Description: Three trocar sites designated as anterior, lateral and posterior were randomized on each patient to receive AZX100 3 mg/cm or AZX100 10 mg/cm or placebo/cm at 9 days and 21 days following shoulder surgery. 3D digital photography of each trocar scar was used to calculate scar length, width, minimum elevation, and maximum elevation in millimeters (mm) at 12 months. The minimum elevation value was calculated as the lowest point of the scar below the interpolated smooth skin surface. This was always a negative number. Negative values (closer to zero) were more desirable. The maximum elevation value was the highest point of the scar above the interpolated smooth skin surface. A smaller value was preferred.
Time Frame: 12 months
Population: Efficacy analysis was based on patient data from the AZX100/Placebo cohort (i.e., not including patients receiving placebo-only). In the ITT sample for the scar objective measures, available sample sizes were 122 at Day 42 and 113 at Month 12 (including four subjects who withdrew from the study but were still followed for safety until Month 12).
Measure: Mean (Standard Deviation); unit: Millimeters
Groups:
- Scar Length for Placebo Trocar Scars: This group included scar length measurements at the 12 month time point for trocar scars that were randomized to receive saline placebo/cm at 9 days and 21 days following shoulder surgery.
- Scar Length for 3 mg AZX100 Trocar Scars: This group included scar length measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 3 mg/cm at 9 days and 21 days following shoulder surgery.
- Scar Length for 10 mg AZX100 Trocar Scars: This group included scar length measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 10 mg/cm at 9 days and 21 days following shoulder surgery.
- Scar Width for Placebo Trocar Scars: This group included scar width measurements at the 12 month time point for trocar scars that were randomized to receive saline placebo/cm at 9 days and 21 days following shoulder surgery.
- Scar Width for 3 mg AZX100 Trocar Scars: This group included scar width measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 3 mg/cm at 9 days and 21 days following shoulder surgery.
- Scar Width for 10 mg AZX100 Trocar Scars: This group included scar width measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 10 mg/cm at 9 days and 21 days following shoulder surgery.
- Scar Minimum Elevation for Placebo Trocar Scars: This group included scar minimum elevation measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 saline placebo/cm at 9 days and 21 days following shoulder surgery.
- Scar Minimum Elevation for 3 mg AZX100 Trocar Scars: This group included scar minimum elevation measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 3 mg/cm at 9 days and 21 days following shoulder surgery.
- Scar Minimum Elevation for 10 mg AZX100 Trocar Scars: This group included scar minimum elevation measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 10 mg/cm at 9 days and 21 days following shoulder surgery.
- Scar Maximum Elevation for Placebo Trocar Scars: This group included scar maximum elevation measurements at the 12 month time point for trocar scars that were randomized to receive saline placebo/cm at 9 days and 21 days following shoulder surgery.
- Scar Maximum Elevation for 3 mg AZX100 Trocar Scars: This group included scar maximum elevation measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 3 mg/cm at 9 days and 21 days following shoulder surgery.
- Scar Maximum Elevation for 10 mg AZX100 Trocar Scars: This group included scar maximum elevation measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 10 mg/cm at 9 days and 21 days following shoulder surgery.
Arm/Group | Scar Length for Placebo Trocar Scars | Scar Length for 3 mg AZX100 Trocar Scars | Scar Length for 10 mg AZX100 Trocar Scars | Scar Width for Placebo Trocar Scars | Scar Width for 3 mg AZX100 Trocar Scars | Scar Width for 10 mg AZX100 Trocar Scars | Scar Minimum Elevation for Placebo Trocar Scars | Scar Minimum Elevation for 3 mg AZX100 Trocar Scars | Scar Minimum Elevation for 10 mg AZX100 Trocar Scars | Scar Maximum Elevation for Placebo Trocar Scars | Scar Maximum Elevation for 3 mg AZX100 Trocar Scars | Scar Maximum Elevation for 10 mg AZX100 Trocar Scars
Number analyzed (Participants) | 113 | 113 | 113 | 113 | 113 | 113 | 113 | 113 | 113 | 113 | 113 | 113
Millimeters | 8.75 (4.12) | 8.74 (3.70) | 9.59 (3.84) | 2.62 (1.50) | 2.59 (1.31) | 2.71 (1.35) | -0.26 (0.19) | -0.29 (0.21) | -0.27 (0.20) | 0.19 (0.17) | 0.18 (0.13) | 0.19 (0.13)
Statistical Analysis 1: Comparison: Scar Length for Placebo Trocar Scars vs Scar Length for 3 mg AZX100 Trocar Scars; Statistical analysis included line plots of paired differences vs. time, univariate p-values from Wilcoxon signed rank tests, and repeated measures regression models in SAS/STAT PROC GENMOD; Test type: Superiority or Other; p = 0.87, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 2: Comparison: Scar Length for Placebo Trocar Scars vs Scar Length for 10 mg AZX100 Trocar Scars; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.15, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 3: Comparison: Scar Width for Placebo Trocar Scars vs Scar Width for 3 mg AZX100 Trocar Scars; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.77, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 4: Comparison: Scar Width for Placebo Trocar Scars vs Scar Width for 10 mg AZX100 Trocar Scars; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.75, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 5: Comparison: Scar Minimum Elevation for Placebo Trocar Scars vs Scar Minimum Elevation for 3 mg AZX100 Trocar Scars; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.050, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 6: Comparison: Scar Minimum Elevation for Placebo Trocar Scars vs Scar Minimum Elevation for 10 mg AZX100 Trocar Scars; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.83, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 7: Comparison: Scar Maximum Elevation for Placebo Trocar Scars vs Scar Maximum Elevation for 3 mg AZX100 Trocar Scars; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.37, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 8: Comparison: Scar Maximum Elevation for Placebo Trocar Scars vs Scar Maximum Elevation for 10 mg AZX100 Trocar Scars; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.43, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used

4. Secondary Outcome: Between-group Mean Differences in Objective Measures Via 3D Photography (Volume)
Description: Three trocar sites designated as anterior, lateral and posterior were randomized on each patient to receive AZX100 3 mg/cm, or AZX100 10 mg/cm, or placebo/cm at 9 days and 21 days following shoulder surgery. 3D digital photography of each trocar scar was used to calculate positive volume, negative volume, and total volume in millimeters cubed (mm^3) at 12 months. Positive volume included the scar volume that was calculated to be above the interpolated smooth skin surface. A smaller value was preferred. Negative volume included the volume of the scar calculated to be below the interpolated smooth skin surface. It was always a negative number; negative values (closer to zero) were more desirable. Total volume was calculated as the sum of positive volume and the absolute value of negative volume. Smaller values were more desirable.
Time Frame: 12 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeters cubed
Groups:
- Scar Positive Volume for Placebo Trocar Scars: This group included scar positive volume measurements at the 12 month time point for trocar scars that were randomized to receive saline placebo/cm at 9 days and 21 days following shoulder surgery.
- Scar Positive Volume for 3 mg AZX100 Trocar Scars: This group included scar positive volume measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 3 mg/cm at 9 days and 21 days following shoulder surgery.
- Scar Positive Volume for 10 mg AZX100 Trocar Scars: This group included scar positive volume measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 10 mg/cm at 9 days and 21 days following shoulder surgery.
- Scar Negative Volume for Placebo Trocar Scars: This group included scar negative volume measurements at the 12 month time point for trocar scars that were randomized to receive saline placebo/cm at 9 days and 21 days following shoulder surgery.
- Scar Negative Volume for 3 mg AZX100 Trocar Scars: This group included scar negative volume measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 3 mg/cm at 9 days and 21 days following shoulder surgery.
- Scar Negative Volume for 10 mg AZX100 Trocar Scars: This group included scar negative volume measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 10 mg/cm at 9 days and 21 days following shoulder surgery.
- Scar Total Volume for Placebo Trocar Scars: This group included scar total volume measurements at the 12 month time point for trocar scars that were randomized to receive saline placebo/cm at 9 days and 21 days following shoulder surgery.
- Scar Total Volume for 3 mg AZX100 Trocar Scars: This group included scar total volume measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 3 mg/cm at 9 days and 21 days following shoulder surgery.
- Scar Total Volume for 10 mg AZX100 Trocar Scars: This group included scar total volume measurements at the 12 month time point for trocar scars that were randomized to receive AZX100 10 mg/cm at 9 days and 21 days following shoulder surgery.
Arm/Group | Scar Positive Volume for Placebo Trocar Scars | Scar Positive Volume for 3 mg AZX100 Trocar Scars | Scar Positive Volume for 10 mg AZX100 Trocar Scars | Scar Negative Volume for Placebo Trocar Scars | Scar Negative Volume for 3 mg AZX100 Trocar Scars | Scar Negative Volume for 10 mg AZX100 Trocar Scars | Scar Total Volume for Placebo Trocar Scars | Scar Total Volume for 3 mg AZX100 Trocar Scars | Scar Total Volume for 10 mg AZX100 Trocar Scars
Number analyzed (Participants) | 113 | 113 | 113 | 113 | 113 | 113 | 113 | 113 | 113
Millimeters cubed | 4.74 (8.95) | 4.05 (4.25) | 4.44 (4.46) | -8.42 (8.66) | -9.44 (12.77) | -9.59 (13.01) | 13.16 (11.53) | 13.49 (13.36) | 14.03 (13.68)
Statistical Analysis 1: Comparison: Scar Positive Volume for Placebo Trocar Scars vs Scar Positive Volume for 3 mg AZX100 Trocar Scars; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.16, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 2: Comparison: Scar Positive Volume for Placebo Trocar Scars vs Scar Positive Volume for 10 mg AZX100 Trocar Scars; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.14, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 3: Comparison: Scar Negative Volume for Placebo Trocar Scars vs Scar Negative Volume for 3 mg AZX100 Trocar Scars; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.69, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 4: Comparison: Scar Negative Volume for Placebo Trocar Scars vs Scar Negative Volume for 10 mg AZX100 Trocar Scars; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.89, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 5: Comparison: Scar Total Volume for Placebo Trocar Scars vs Scar Total Volume for 3 mg AZX100 Trocar Scars; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.30, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 6: Comparison: Scar Total Volume for Placebo Trocar Scars vs Scar Total Volume for 10 mg AZX100 Trocar Scars; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.46, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used

5. Secondary Outcome: Histological Evaluation of Collagen
Description: Three trocar sites designated as anterior, lateral and posterior were randomized on each patient to receive AZX100 3 mg/cm or AZX100 10 mg/cm or placebo/cm at 9 days and 21 days following shoulder surgery. A skin punch biopsy was taken of each trocar site at 12 months. The specimens were blindly scored in duplicate by a dermal pathologist for dermal collagen fiber density, maturity and orientation, where 0% was completely normal and 100% was completely abnormal.
Time Frame: 12 months
Population: This analysis was based on patient data from the AZX100/Placebo cohort (i.e., not including patients receiving placebo-only). In the ITT sample for the histology analyses, available sample sizes were 122 at Day 42 and 113 at Month 12 (including four subjects who withdrew from the study but were still followed for safety until Month 12).
Measure: Mean (Standard Deviation); unit: Percent
Groups:
- Collagen Fiber Density Results for Placebo Scars: This group included results for collagen fiber density at the 12 month time point for trocar scars that were randomized to receive saline placebo/cm at 9 days and 21 days following shoulder surgery.
- Collagen Fiber Density Results for 3 mg AZX100 Scars: This group included results for collagen fiber density at the 12 month time point for trocar scars that were randomized to receive AZX100 3 mg/cm at 9 days and 21 days following shoulder surgery.
- Collagen Fiber Density Results for 10 mg AZX100 Scars: This group included results for collagen fiber density at the 12 month time point for trocar scars that were randomized to receive AZX100 10 mg/cm at 9 days and 21 days following shoulder surgery.
- Collagen Fiber Maturity Results for Placebo Scars: This group included results for collagen fiber maturity at the 12 month time point for trocar scars that were randomized to receive saline placebo/cm at 9 days and 21 days following shoulder surgery.
- Collagen Fiber Maturity Results for 3 mg AZX100 Scars: This group included results for collagen fiber maturity at the 12 month time point for trocar scars that were randomized to receive AZX100 3 mg/cm at 9 days and 21 days following shoulder surgery.
- Collagen Fiber Maturity Results for 10 mg AZX100 Scars: This group included results for collagen fiber maturity at the 12 month time point for trocar scars that were randomized to receive AZX100 10 mg/cm at 9 days and 21 days following shoulder surgery.
- Collagen Fiber Orientation Results for Placebo Scars: This group included results for collagen fiber orientation at the 12 month time point for trocar scars that were randomized to receive saline placebo/cm at 9 days and 21 days following shoulder surgery.
- Collagen Fiber Orientation Results for 3 mg AZX100 Scars: This group included results for collagen fiber orientation at the 12 month time point for trocar scars that were randomized to receive AZX100 3 mg/cm at 9 days and 21 days following shoulder surgery.
- Collagen Fiber Orientation Results for 10 mg AZX100 Scars: This group included results for collagen fiber orientation at the 12 month time point for trocar scars that were randomized to receive AZX100 10 mg/cm at 9 days and 21 days following shoulder surgery.
Arm/Group | Collagen Fiber Density Results for Placebo Scars | Collagen Fiber Density Results for 3 mg AZX100 Scars | Collagen Fiber Density Results for 10 mg AZX100 Scars | Collagen Fiber Maturity Results for Placebo Scars | Collagen Fiber Maturity Results for 3 mg AZX100 Scars | Collagen Fiber Maturity Results for 10 mg AZX100 Scars | Collagen Fiber Orientation Results for Placebo Scars | Collagen Fiber Orientation Results for 3 mg AZX100 Scars | Collagen Fiber Orientation Results for 10 mg AZX100 Scars
Number analyzed (Participants) | 113 | 113 | 113 | 113 | 113 | 113 | 113 | 113 | 113
Percent | 24.20 (24.08) | 19.43 (21.79) | 25.34 (23.18) | 22.72 (23.59) | 17.95 (21.52) | 23.64 (22.68) | 23.41 (24.54) | 18.52 (21.73) | 24.77 (24.00)
Statistical Analysis 1: Comparison: Collagen Fiber Density Results for Placebo Scars vs Collagen Fiber Density Results for 3 mg AZX100 Scars; Agreement between the two rater evaluations was assessed by tabulating the difference of the two ratings. Statistical methods for paired data were used to compare the two dosages of AZX100 to placebo; Test type: Superiority or Other; p = 0.086, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 2: Comparison: Collagen Fiber Density Results for Placebo Scars vs Collagen Fiber Density Results for 10 mg AZX100 Scars; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.66, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 3: Comparison: Collagen Fiber Maturity Results for Placebo Scars vs Collagen Fiber Maturity Results for 3 mg AZX100 Scars; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.069, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 4: Comparison: Collagen Fiber Maturity Results for Placebo Scars vs Collagen Fiber Maturity Results for 10 mg AZX100 Scars; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.68, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 5: Comparison: Collagen Fiber Orientation Results for Placebo Scars vs Collagen Fiber Orientation Results for 3 mg AZX100 Scars; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.095, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used
Statistical Analysis 6: Comparison: Collagen Fiber Orientation Results for Placebo Scars vs Collagen Fiber Orientation Results for 10 mg AZX100 Scars; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.62, Wilcoxon (signed rank) — For this early phase study, multiple comparisons adjustments were not used

6. Secondary Outcome: Histological Evaluation of Number of Alpha Smooth Muscle Actin Cells
Description: Three trocar sites designated as anterior, lateral and posterior were randomized on each patient to receive AZX100 3 mg/cm or AZX100 10 mg/cm or placebo/cm at 9 days and 21 days following shoulder surgery. A skin punch biopsy was taken of each trocar site at 12 months. For exploratory purposes, the specimens were blindly scored in duplicate by a dermal pathologist for the estimated number of alpha-smooth muscle actin (α-SMA) positive cells per high powered field. Values ranged from 0 to several hundred. The number of α-SMA cells was assessed for exploratory purposes; therefore, at the time of this report, it was not known whether it was better to have a low or high α-SMA score.
Time Frame: 12 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Cells per high-powered field
Groups:
- Alpha SMA Results for Placebo Trocar Scars: This group included assessment for α-SMA at the 12 month time point for trocar scars that were randomized to receive saline placebo/cm at 9 days and 21 days following shoulder surgery.
- Alpha SMA Results for 3 mg AZX100 Trocar Scars: This group included assessment for α-SMA at the 12 month time point for trocar scars that were randomized to receive AZX100 3 mg/cm at 9 days and 21 days following shoulder surgery.
- Alpha SMA Results for 10 mg AZX100 Trocar Scars: This group included assessment for α-SMA at the 12 month time point for trocar scars that were randomized to receive AZX100 10 mg/cm at 9 days and 21 days following shoulder surgery.
Arm/Group | Alpha SMA Results for Placebo Trocar Scars | Alpha SMA Results for 3 mg AZX100 Trocar Scars | Alpha SMA Results for 10 mg AZX100 Trocar Scars
Number analyzed (Participants) | 113 | 113 | 113
Cells per high-powered field | 22.07 (47.02) | 24.78 (58.25) | 32.80 (64.56)
Statistical Analysis 1: Comparison: Alpha SMA Results for Placebo Trocar Scars vs Alpha SMA Results for 3 mg AZX100 Trocar Scars; A regression analysis was run to compare alpha-SMA between 3 mg and 10 mg AZX100 and placebo, adjusted for the subject's gender and age. GEE regression in SAS/STAT PROC GENMOD was used because it properly handled the correlations among the three observations for each subject; Test type: Superiority or Other; p = 0.44, Wilcoxon (signed rank)
Statistical Analysis 2: Comparison: Alpha SMA Results for Placebo Trocar Scars vs Alpha SMA Results for 10 mg AZX100 Trocar Scars; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.41, Wilcoxon (signed rank)

ADVERSE EVENTS:
Time Frame: Adverse events began to be collected for each patient after dosing with study agent, and were collected for the duration of the study (12 months). The adverse event collection period for the entire study lasted for a period of 24 months.
Description: All 150 treated subjects were included in the adverse event analyses. Two groups were compared: 126 subjects who received placebo, 3 mg/cm, and 10 mg/cm of AZX100 at three shoulder trocar sites; and 24 subjects who received only placebo at three shoulder trocar sites.
Arm/Group | AZX100-Placebo Arm | Placebo-only Arm
Serious Adverse Events (participants affected / at risk) | 8/126 | 2/24
Other Adverse Events (participants affected / at risk) | 125/126 | 21/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZX100-Placebo Arm (N=126) | Placebo-only Arm (N=24)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 1 (1)
Cholecystitis, Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Coronary Artery Occlusion (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Transient Ischemic Attack (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZX100-Placebo Arm (N=126) | Placebo-only Arm (N=24)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 1 (1)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 4 (4)
Dizziness (Nervous system disorders) | 7 (7) | 2 (3)
Fatigue (General disorders) | 0 (0) | 2 (4)
Headache (Nervous system disorders) | 7 (7) | 3 (6)
Influenza (Infections and infestations) | 2 (2) | 3 (3)
Injection Site Erythema (General disorders) | 46 (106) | 3 (5) — Special note for injection site adverse events: There were three trocar treatment areas on the shoulder; therefore, a participant could have the same and/or different injection site events at all three trocar treatment sites simultaneously.
Injection Site Irritation (General disorders) | 63 (163) | 6 (15) — Special note for injection site adverse events: There were three trocar treatment areas on the shoulder; therefore, a participant could have the same and/or different injection site events at all three trocar treatment sites simultaneously.
Injection Site Pain (General disorders) | 80 (246) | 7 (23) — Special note for injection site adverse events: There were three trocar treatment areas on the shoulder; therefore, a participant could have the same and/or different injection site events at all three trocar treatment sites simultaneously.
Injection Site Pruritus (General disorders) | 14 (21) | 2 (5) — Special note for injection site adverse events: There were three trocar treatment areas on the shoulder; therefore, a participant could have the same and/or different injection site events at all three trocar treatment sites simultaneously.
Injection Site Urticaria (General disorders) | 24 (61) | 1 (3) — Special note for injection site adverse events: There were three trocar treatment areas on the shoulder; therefore, a participant could have the same and/or different injection site events at all three trocar treatment sites simultaneously.
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 12 (17) | 2 (4)
Nasopharyngitis (Infections and infestations) | 8 (8) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (8) | 1 (1)
Oedema Peripheral (General disorders) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 10 (12) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 19 (26) | 6 (6)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less